CLINICAL TRIAL: NCT04745637
Title: Managed Access Programs for INC424, Ruxolitinib
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424A2405
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Primary Myelofibrosis (PMF); Post Polycythemia Myelofibrosis (PPV MF); Thrombocythemia Myelofibrosis (PET-MF); Severe/Very Severe COVID-19 Illness; Polycythemia Vera (PV); Steroid Refractory Acute Graft Versus Host Disease (SR aGVHD); Steroid Refractory Chronic Graft Versus Host Disease (SR cGVHD)
Keywords: MAP; Manage Access Program; Primary Myelofibrosis (PMF); Post Polycythemia Myelofibrosis (PPV MF); Thrombocythemia Myelofibrosis (PET-MF); Severe/very severe COVID-19 illness; Polycythemia Vera (PV); Steroid refractory acute Graft versus Host Disease (SR aGVHD); Steroid refractory chronic Graft versus Host Disease (SR cGVHD); INC424; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ruxolitinib — Patients receive Ruxolitinib
  Other Names: INC424

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to INC424, Ruxolitinib

DETAILED DESCRIPTION:
CINC424A2405 - No longer available- Managed Access Program (MAP) Cohort Treatment Plan CINC424A2405 to provide access to Ruxolitinib for patients with Primary Myelofibrosis (PMF) or Post Polycythemia Myelofibrosis (PPV MF) or Post-Essential Thrombocythemia Myelofibrosis (PET-MF)

CINC424A2001M - No longer available - Ruxolitinib Managed Access Program (MAP) for patients diagnosed with severe/very severe COVID-19 illness

CINC424B2002I - No longer available- Managed Access Program (MAP) Cohort Treatment Plan CINC424B2002I to provide access to Ruxolitinib for patients with Polycythemia Vera (PV)

CINC424C2001M - Available - Managed Access Program (MAP) Cohort Treatment Plan CINC424C2001M to provide access to ruxolitinib for steroid refractory acute and chronic Graft versus Host Disease (SR aGVHD and SR cGHVD).

ELIGIBILITY:
Inclusion criteria

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enroll in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult